CLINICAL TRIAL: NCT06320938
Title: Comparison of the Effects of Neuroscience-Based Pain Education and Myofascial Induction Technique on Pain and Quality of Life in Patients With Chronic Neck Pain
Brief Title: Effectiveness of Neuroscience-based Pain Education in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkoglu Dr. Kemal Beyazit State Hospital (Other)
Responsible Party: Principal Investigator, Süreyya DAMAR ÖRENLER, Principal Investigator, Turkoglu Dr. Kemal Beyazit State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/18
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-08

CONDITIONS: Cervical Spine Disease
Keywords: Pain neuroscience education; Myofascial induction technique; Myofascial treatment; Home exercises; Pain; Neck Disability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuroscience-Based Pain Education Combined with Home Exercise Program (Active Comparator): Patients in this group will receive Neuroscience-Based Pain Education (NPE) treatment in addition to the home exercise program. Training sessions are planned once a week for an average of 35-45 minutes and 8 sessions. NPE will be performed by a physiotherapist who has an internationally recognized certificate in this regard. Training sessions will be organized as one-on-one conversation sessions focusing on the neurophysiology of pain, and patients will be reinforced through PowerPoint presentations and visual pictures, templates, and metaphors.
  Interventions: Other: Neuroscience-Based Pain Education Combined with Home Exercise Program
- Myofascial Induction Techniques Combined with Home Exercise Program (Active Comparator): In addition to the home exercise program, Myofascial Induction Techniques (MIT) group patients will have MIT applied to the cervical and upper thoracic regions by a physiotherapist trained and experienced in myofascial treatments. The application will be once a week for 8 weeks, with an average duration of 35-45 minutes.
  Interventions: Other: Myofascial Induction Techniques Combined with Home Exercise Program
- Home Exercise Program (Active Comparator): Patients in this group will be taught an exercise program after undergoing general training. Exercises will include stretching and strengthening exercises for neck muscles and posture exercises. Patients are asked to take 35-45 minutes once a day, five days a week, for 8 weeks. They will be asked to do the given home exercises and fill out follow-up charts. The continuity of the exercises will be ensured by sending reminder messages to this group of patients once a week by the physiotherapist about doing their exercises.
  Interventions: Other: Home Exercises Group

INTERVENTIONS:
Other: Neuroscience-Based Pain Education Combined with Home Exercise Program — Neuroscience-Based Pain Education and Home Exercises will be applied.
  Arms: Neuroscience-Based Pain Education Combined with Home Exercise Program
Other: Myofascial Induction Techniques Combined with Home Exercise Program — Myofascial Induction Techniques and Home Exercises will be applied.
  Arms: Myofascial Induction Techniques Combined with Home Exercise Program
Other: Home Exercises Group — Home Exercises wiil be applied
  Arms: Home Exercise Program

SUMMARY:
The effectiveness of neuroscience-based pain education, myofascial induction technique, and home exercise programs will be compared in patients with chronic neck pain.

DETAILED DESCRIPTION:
The study aims to present the immediate and long-term effects of Neuroscience-based Pain Education (NPE) and Myofascial Induction Therapy (MIT). It will evaluate parameters such as pain, quality of life, pain catastrophizing, and neck disability after treatment completion and at the 6-month follow-up.

The investigators aim to illuminate future studies concerning neuroscience-based pain education, which has gained prominence in recent years and continues to increase in importance annually.

The participants will be randomly assigned to one of three groups:

1 Group: Neuroscience-Based Pain Education Combined with Home Exercise Program Participants in this group will receive Neuroscience-Based Pain Education (NPE) treatment in addition to the home exercise program. Training sessions will be organized as one-on-one conversation sessions focusing on the neurophysiology of pain, and participants will be reinforced through PowerPoint presentations and visual aids such as pictures, templates, and metaphors.

Group: Myofascial Induction Techniques Combined with Home Exercise Program In addition to the home exercise program, Myofascial Induction Techniques (MIT) group participants will have MIT applied to the cervical and upper thoracic regions.

Group: Home Exercise Program After undergoing general training, participants in this group will be taught an exercise program. The program will include neck muscle stretching, strengthening, and posture exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18-60 years old,
2. Patients with non-specific neck pain for at least 3 months,
3. Having pain severity of four or more according to the Visual analogue scale (VAS),
4. Patients with Pain Catastrophizing Scale score > 30
5. Patients with a Central Sensitization Inventory score > 30
6. Not having received physiotherapy and manual therapy within the last 3 months,
7. Those who have not received and will not receive medical treatment in the last 3 months.

Exclusion Criteria:

1. Having a history of neck and spine surgery,
2. Patients with whiplash injury, fracture history,
3. Having unstable neurological findings,
4. Presence of a pathology such as hernia and root compression in the cervical region,
5. Those who regularly use analgesic and anti-inflammatory drugs,
6. A communication problem may prevent the implementation of the evaluations or treatment program.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Short Form McGill Pain Questionnaire | Baseline,8 weeks, 6 months
  A short form of the McGill Pain Questionnaire (SF-MPQ) used in pain assessment consists of four sections. In the first section, participants are asked to mark the location of pain on a body diagram. In the second section, participants are asked to select the word that best describes their pain from twenty subgroups. The third section investigates the relationship of pain over time, while the fourth and final section requires participants to indicate the intensity of pain on a scale of 1 to 5 and provide written responses to six questions. The questionnaire is scored from 0 to 112. The higher the pain score, the greater the pain.
Algometric Digital Measurement | Baseline,8 weeks, 6 months
  It is a digital device used to evaluate trigger point sensitivity.
Central Sensitization Inventory | Baseline,8 weeks, 6 months
  The scale, which can be applied in chronic pain, is used in central sensitization syndromes. It consists of two parts. Section A questions health-related symptoms, and part B questions whether any central sensitization syndromes have been diagnosed before.
Head Posture Evaluation | Baseline,8 weeks, 6 months
  Forward head posture is measured with a goniometer, which measures the angle between the horizontal plane and the seventh cervical vertebra and ear line.
Neck Disability Index | Baseline,8 weeks, 6 months
  The scale consists of ten headings in total. It includes neck pain intensity, personal care, lifting, reading, headaches, concentration, driving, sleep, and leisure activities.
Pittsburgh Sleep Quality Index | Baseline,8 weeks, 6 months
  This survey contains 24 questions about sleep status, both during the day and at night. Nineteen of these are to be answered personally, and five are to be answered by a spouse or roommate.
36-Item Short Form Health Survey Questionnaire | Baseline,8 weeks, 6 months
  36-Item Short Form Health Survey (SF-36) questionnaire consists of eight subscales: physical functioning, social functioning, role limitations due to physical problems, pain, vitality, mental health, and general health perception. Each subscale is scored from 0 to 100, and the scores from these subscales are not summed. A high score indicates good health status.
Pain Catastrophizing Scale | Baseline,8 weeks, 6 months
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure of catastrophizing in the context of actual or anticipated pain. The PCS measures catastrophizing as a multidimensional construct with three subscales: rumination, magnification, and helplessness. Rumination focuses on thoughts related to pain, helplessness reflects feelings of helplessness in coping with a painful situation, and magnification is a general view of the threat of pain. High PCS scores are associated with greater pain and more functional impairment. A total score above 30 represents clinically significant levels of pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, Assoc. Prof., Study Director — Hasan Kalyoncu University
Locations (1):
- Türkoğlu Dr. Kemal Beyazıt State Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernetti A, Agostini F, de Sire A, Mangone M, Tognolo L, Di Cesare A, Ruiu P, Paolucci T, Invernizzi M, Paoloni M. Neuropathic Pain and Rehabilitation: A Systematic Review of International Guidelines. Diagnostics (Basel). 2021 Jan 5;11(1):74. doi: 10.3390/diagnostics11010074. PMID 33466426
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Javdaneh N, Saeterbakken AH, Shams A, Barati AH. Pain Neuroscience Education Combined with Therapeutic Exercises Provides Added Benefit in the Treatment of Chronic Neck Pain. Int J Environ Res Public Health. 2021 Aug 22;18(16):8848. doi: 10.3390/ijerph18168848. PMID 34444594